CLINICAL TRIAL: NCT04954794
Title: A Phase II Study of Transcatheter Arterial Chemoembolization (TACE) Combined with Sintilimab Plus Bevacizumab Biosimilar in Patients with Advanced Hepatocellular Carcinoma (TASK-02)
Brief Title: TACE Combined with Sintilimab Plus Bevacizumab Biosimilar in Patients with Advanced Hepatocellular Carcinoma (TASK-02)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Peng Wang, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIT-011
Record Dates: First submitted 2021-07-01; First posted 2021-07-08 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TACE in combination with Sintilimab plus a bevacizumab biosimilar (Experimental)
  Interventions: Drug: Sintilimab; Combination Product: TACE

INTERVENTIONS:
Drug: Sintilimab — Sintilimab will be administered at 200 mg i.v. every 3 weeks plus a bevacizumab biosimilar at 15 mg/kg i.v. every 3 weeks until documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
Combination Product: TACE — TACE is performed by using drug-eluting beads or using microspheres combined with Lipiodol-pirarubicin emulsion per Investigator's decision. TACE treatment starts at day 0. Sintilimab plus a bevacizumab biosimilar will be initiated on day 14 after TACE.

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of TACE combined with Sintilimab plus bevacizumab biosimilar in patients with advanced hepatocellular carcinoma as first-line therapy.

DETAILED DESCRIPTION:
Transarterial chemoembolization (TACE) is commonly used for the treatment of advanced hepatocellular carcinoma. Early randomized trials suggested that TACE can be accepted as the standard treatment for advanced-stage disease. However, the outcome of patients treated with TACE in real-life cohorts is still very poor.

Recent studies have also supported a safe combination of immune checkpoint inhibition with TACE. And the combination of sintilimab plus bevacizumab biosimilar showed significantly improved survival in advanced HCC. Therefore, the objective of this study is to evaluate the efficacy and safety of TACE combined with anti-PD-1 antibody in patients in advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained.
* Age ≥ 18 years at time of study entry.
* Barcelona Clinic Liver Cancer stage C.
* Histologically confirmed diagnosis of HCC.
* At least one measurable site of disease as defined by RECIST1.1criteria with spiral CT scan or MRI，apart from one liver lesion to serve for TACE.
* Child-Pugh scores 5-7, performance status (PS) ≤ 2 (ECOG scale).
* Subjects with chronic HBV infection must have HBV DNA viral load < 100 IU/mL at screening. In addition, they must be on antiviral therapy per regional standard of care guidelines prior to initiation of study therapy.
* Life expectancy of at least 12 weeks.
* Adequate blood count, liver-enzymes, and renal function: absolute neutrophil count ≥ 1,500/L, platelets ≥60 x103/L; Total bilirubin ≤ 3x upper normal limit; Aspartate Aminotransferase (SGOT), Alanine aminotransferase (SGPT) ≤ 5 x upper normal limit (ULN); International normalized ratio (INR) ≤1.25; Albumin ≥ 31 g/dL; Serum Creatinine ≤ 1.5 x institutional ULN or creatinine clearance (CrCl) ≥ 30 mL/min (if using the Cockcroft-Gault formula)
* Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment, adherence to contraceptive measures, scheduled visits and examinations including follow up.

Exclusion Criteria:

* Patients on a liver transplantation list or with advanced liver disease.
* Total thrombosis or total invasion of the main branch of the portal vein.
* History of cardiac disease, including clinically significant gastrointestinal bleeding within 4 weeks prior to start of study treatment
* Thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months Prior to the first dose of study drug with the exception of thrombosis of a segmental portal vein.
* Prior systemic anti-cancer therapy OR endocrine- OR immunotherapy
* Prior treatment with TACE
* RFA and resection administered less then 4 weeks prior to study treatment start.
* Radiotherapy administered less then 4 weeks prior to study treatment start.
* Major surgery within 4 weeks of starting the study treatment OR subjects who have not recovered from effects of major surgery.
* Patients with second primary cancer, except adequately treated basal skin cancer or carcinoma in-situ of the cervix.
* Immunocompromised patients, e.g. patients who are known to be serologically positive for human immunodeficiency virus (HIV).
* Participation in another clinical study with an investigational product during the last 30 days before inclusion or 7 half-lifes of previously used trial medication, whichever is longer.
* Previous treatment in the present study (does not include screening failure).
* Any condition or comorbidity that, in the opinion of the investigator, would interfere with evaluation of study Treatment or interpretation of patient safety or study results, including but not limited to:

  1. history of interstitial lung disease
  2. Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) coinfection (i.e double infection)
  3. known acute or chronic pancreatitis
  4. active tuberculosis
  5. any other active infection (viral, fungal or bacterial) requiring systemic therapy
  6. history of allogeneic tissue/solid organ transplant
  7. diagnosis of immunodeficiency or patient is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of nivolumab-monotherapy treatment.
  8. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Exceptions: Subjects with vitiligo, hypothyroidism, diabetes mellitus type I or resolved childhood asthma/atopy are an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with Hashimoto thyroiditis, hypothyroidism stable on hormone replacement or psoriasis not requiring treatment are not excluded from the study.
  9. Live vaccine within 30 days prior to the first dose of nivolumab-monotherapy treatment or during study treatment.
  10. History or clinical evidence of Central Nervous System (CNS) metastases Exceptions are: Subjects who have completed local therapy and who meet both of the following criteria: I. are asymptomatic and II. have no requirement for steroids 6 weeks prior to start of nivolumab-monotherapy treatment. Screening with CNS imaging (CT or MRI) is required only if clinically indicated or if the subject has a history of CNS.
* Medication that is known to interfere with any of the agents applied in the trial.
* Any other efficacious cancer treatment except protocol specified treatment at study start.
* Patient has received any other investigational product within 28 days of study entry.
* Prior therapy with an anti-Programmed cell death protein 1 (anti-PD-1), anti-PD-L1, anti-Programmed cell death-ligand 2 (anti-PD-L2), anti-CD137 (4-1BB ligand, a member of the Tumor Necrosis Factor Receptor (TNFR) family), or anti-Cytotoxic T-lymphocyte-associated antigen-4 (anti-CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Female subjects who are pregnant, breast-feeding or male/female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year). [Acceptable methods of contraception are: implants, injectable contraceptives, combined oral contraceptives, intrauterine pessars (only hormonal devices), sexual abstinence or vasectomy of the partner]. Women of childbearing potential must have a negative pregnancy test (serum β-HCG) at screening.
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | max 24 months
  ORR according to RECIST 1.1 for HCC

SECONDARY OUTCOMES:
Duration of Response | max 24 months
Progression-Free Survival | max 24 months
Overall survival | max 42 months
Disease control rate | max 24 months
Adverse Events | max 42 months
  Adverse event (AE)、Treatment emergent adverse event(TEAE)、Serious adverse event (SAE).

CONTACTS AND LOCATIONS:
Overall Officials: Peng Wang, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No